CLINICAL TRIAL: NCT02519062
Title: FDG-PET, Marker Immunologici ed Ipossici in Pazienti Affetti da Carcinoma Polmonare Non a Piccole Cellule in Stadio I-III Sottoposti a Chirurgia Radicale
Brief Title: Role of FDG PET, Immune and Hypoxic Marker in NSCLC
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1332
Record Dates: First submitted 2015-06-26; First posted 2015-08-10 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma; Non-Small-Cell Lung; FDG PET; hypoxia markers; immune markers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tumor surgical specimen
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This is a retrospective study

SUMMARY:
This is a retrospective study that involves the revision of clinical, instrumental and pathologic data of an estimated cohort of maximum 130 patients with NSCLC treated with surgery with radical intent at our center.

DETAILED DESCRIPTION:
This is a retrospective observation that involves the revision of clinical, instrumental and pathologic data of an estimated cohort of 130 patients with NSCLC treated with surgery with radical intent at our center.

We will review FDG-PET acquired within 30 days prior to surgery and analyze its principal imaging characteristics with respect to hypoxic and immune-related markers at immunohistochemistry (IHC). These markers will be studied on tumor tissue obtained at surgery, used for diagnostic purposes and stored in paraffin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSCLC (Stage I-III)
* FDG PET before surgery

Exclusion Criteria:

* Absence of tumor specimen
* No clinical data
* FDG-PET can not be evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit a maximum number of 130 NSCLC patients operated radically (stage I-III) at our institution during 2010-2014, of which are available clinical and instrumental data and surgical tumor specimen.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Correlation of SUVmax (Maximal Standardized Uptake Value) in patients with non-small cell lung cancer undergoing surgery with hypoxia expression and tumor immune cell infiltration. | Baseline SUVmax up to 1 month before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Egesta Lopci, MD, Principal Investigator — Humanitas Clinical and Research Hospital
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Background] Lopci E, Grassi I, Chiti A, Nanni C, Cicoria G, Toschi L, Fonti C, Lodi F, Mattioli S, Fanti S. PET radiopharmaceuticals for imaging of tumor hypoxia: a review of the evidence. Am J Nucl Med Mol Imaging. 2014 Jun 7;4(4):365-84. eCollection 2014. PMID 24982822
- [Background] Saintigny P, Burger JA. Recent advances in non-small cell lung cancer biology and clinical management. Discov Med. 2012 Apr;13(71):287-97. PMID 22541616
- [Background] Vaupel P, Mayer A. Hypoxia in cancer: significance and impact on clinical outcome. Cancer Metastasis Rev. 2007 Jun;26(2):225-39. doi: 10.1007/s10555-007-9055-1. PMID 17440684
- [Background] Lopci E, Toschi L, Grizzi F, Rahal D, Olivari L, Castino GF, Marchetti S, Cortese N, Qehajaj D, Pistillo D, Alloisio M, Roncalli M, Allavena P, Santoro A, Marchesi F, Chiti A. Correlation of metabolic information on FDG-PET with tissue expression of immune markers in patients with non-small cell lung cancer (NSCLC) who are candidates for upfront surgery. Eur J Nucl Med Mol Imaging. 2016 Oct;43(11):1954-61. doi: 10.1007/s00259-016-3425-2. Epub 2016 Jun 1. PMID 27251642
- [Background] Castello A, Grizzi F, Toschi L, Rossi S, Rahal D, Marchesi F, Russo C, Finocchiaro G, Lopci E. Tumor heterogeneity, hypoxia, and immune markers in surgically resected non-small-cell lung cancer. Nucl Med Commun. 2018 Jul;39(7):636-644. doi: 10.1097/MNM.0000000000000832. PMID 29608508
- [Background] Grizzi F, Castello A, Qehajaj D, Toschi L, Rossi S, Pistillo D, Paleari V, Veronesi G, Novellis P, Monterisi S, Mineri R, Rahal D, Lopci E. Independent expression of circulating and tissue levels of PD-L1: correlation of clusters with tumor metabolism and outcome in patients with non-small cell lung cancer. Cancer Immunol Immunother. 2019 Sep;68(9):1537-1545. doi: 10.1007/s00262-019-02387-9. Epub 2019 Sep 3. PMID 31482306
- [Background] Grizzi F, Castello A, Qehajaj D, Russo C, Lopci E. The Complexity and Fractal Geometry of Nuclear Medicine Images. Mol Imaging Biol. 2019 Jun;21(3):401-409. doi: 10.1007/s11307-018-1236-5. PMID 30003453